CLINICAL TRIAL: NCT07051837
Title: Background: Isometric Handgrip (IHG) is a Classic Sympatho- Excitatory Stimulus Often Used in Autonomic Testing. Aims: The Aims of This Study Were to Evaluate the Acute Cardiovascular Response and Recovery Following Isometric Handgrip (HG) Exercise-induced Fatigue on Healthy Adults. Secondary, to Examine Correlations Between Isometric Handgrip Strength and Both Systolic (SBP) and Diastolic (DPB) Blood Pressure' Methods: Study Was a Repeated Measure Single Group Design. Thirty-five Healthy Volunteers, 20 Females and 15 Males, Age (36.16 + 6.11years) Were Enrolled in the Study. Study Was at Out
Brief Title: Background: Isometric Handgrip (IHG) is a Classic Sympatho- Excitatory Stimulus Often Used in Autonomic Testing. Aims: The Aims of This Study Were to Evaluate the Acute Cardiovascular Response and Recovery Following Isometric Handgrip (HG) Exercise-induced Fatigue on Healthy Adults. Secondary, to e
Status: Completed | Type: Observational
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Amira Mohamed Afify, ASSOCIATE PROFESSOR OF 1Department of Physical Therapy for Cardiopulmonary Disorders and Geriatrics, Faculty of Physical Therapy, October 6 University
Other Study IDs: P.T.REC/012/005645
Record Dates: First submitted 2025-06-24; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Isometric Exercise

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
: Isometric handgrip (IHG) is a classic sympatho- excitatory stimulus often used in autonomic testing.

Aims: The aims of this study were to evaluate the acute cardiovascular response and recovery following isometric handgrip (HG) exercise-induced fatigue on healthy adults. Secondary, to examine correlations between isometric handgrip strength and both systolic (SBP) and diastolic (DPB) blood pressure' Methods: Study was a repeated measure single group design. Thirty-five healthy volunteers, 20 females and 15 males, age (36.16 + 6.11years) were enrolled in the study. Study was at out Clinic of October 6 University. Demographic data were collected at beginning of session. Subjects were then assessed for baseline (BL) blood pressure (BP). Maximal isometric voluntary contraction (MIVC) for each subject was the average of two-5 seconds MIVCs of dominant hand using a hand-held dynamometer separated by 1 minute of rest. Subjects were allowed 5 minutes rest, then performed fatigue protocol (FP) using the hand-held dynamometer with their dominant hand at 50% MIVC for 3 minutes as a One minute of rest was given following FP then subjects were reassessed for BP and MIVC of dominant hand respectively (Immediate reassessment). Further, BP was reassessed for 3 times at 5 minutes interval between measures.

ELIGIBILITY:
Inclusion Criteria:

* Participants should fulfil the criteria set for age and BMI ranges. All participants should be medically stable and normotensive. They should not have any physical limitations that prevent performance of IHG exercises.

Exclusion Criteria:

* Patients will be excluded from the study if they are smokers, under any medications, diabetics, diagnosed with cardiovascular diseases. Also if they have orthopaedic limitations or mental problems that affect the participation and the result of the study

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Thirty-five healthy participants will be recruited to conduct this study. Their age will range between 20 and 40 years, and body mass index (BMI) between 25- 29.9 kg/m2.
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2024-04-02 (Actual); Primary Completion 2025-04-03 (Actual); Study Completion 2025-05-06 (Actual)

PRIMARY OUTCOMES:
to evaluate the acute cardiovascular response and recovery following isometric handgrip exercise-induced fatigue on healthy adults. and to examine correlations between isometric handgrip strength and both systolic and diastolic blood pressure | from April 2024toMay 2025
  Maximal isometric voluntary contraction (MIVC) for each subject was the average of two-5 seconds MIVCs of dominant hand using a hand-held dynamometer separated by 1 minute of rest. Subjects were allowed 5 minutes rest, then performed fatigue protocol (FP) using the hand-held dynamometer with their dominant hand at 50% MIVC for 3 minutes as a One minute of rest was given following FP then subjects were reassessed for BP and MIVC of dominant hand respectively (Immediate reassessment). Further, BP was reassessed for 3 times at 5 minutes interval between measures

CONTACTS AND LOCATIONS:
Locations (1):
- Amira Mohamed Afify, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No